CLINICAL TRIAL: NCT02717052
Title: Positron Emission Tomography Assessment of Ketamine Binding of the Serotonin Transporter and Its Relevance for Rapid Antidepressant Response
Brief Title: Positron Emission Tomography Assessment of Ketamine Binding of the Serotonin Transporter
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Lanzenberger, Assoc. Prof. PD Dr. Rupert Lanzenberger, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1643/2014; 2014-003280-38 (EudraCT Number)
Record Dates: First submitted 2016-03-11; First posted 2016-03-23 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Depression; Ketamine
MeSH Terms: conditions — Depression | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Pilot I and Pilot III not randomised
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- (S)-ketamine (Experimental): Ketanest® S (Esketaminhydrochlorid) 5mg/ml and 25mg/ml ampoules; Actavis Italy S.P.A./Pfizer Corporation Austria GmbH
  Dosis: 0.25mg/kg bodyweight i.v. over 40 Minutes (ending 10 minutes before PET measurement)
  all patients and 10 HC (randomized, double blind)
  Interventions:
  Drug: (S)-ketamine (Main study) Other: Main study: PET1 Other: Main study: PET2
  Interventions: Drug: (S)-ketamine (Main study); Other: Main Study: PET1; Other: Main Study: PET2
- Placebo (Placebo Comparator): 0.9% saline solution i.v. over 40 Minutes (ending 10 minutes before PET measurement)
  10 HC (randomized, double blind)
  Interventions:
  Drug: Placebo Other: Main study: PET1 Other: Main study: PET2
  Interventions: Drug: Placebo; Other: Main Study: PET1; Other: Main Study: PET2
- (S)-ketamine (Pilot Study II, 5 subj.) (Experimental): Ketanest® S (Esketaminhydrochlorid) 5mg/ml and 25mg/ml ampoules; Actavis Italy S.P.A./Pfizer Corporation Austria GmbH
  Dosis: 0.10mg/kg bodyweight bolus applied over 5 minutes (starting 15 minutes before PET measurement) and continuous infusion of 0.30mg/kg bodyweight applied over the course of 130 minutes.
  Pilot-study II is cross-over design!
  Interventions:
  Drug: (S)-ketamine (Pilot II) Other: PILOT Study II: PET1 Other: PILOT Study II: PET2
  Interventions: Drug: (S)-ketamine (Pilot II); Other: PILOT Study II: PET1; Other: PILOT Study II: PET2
- (R,S)-ketamine (Pilot Study II, 5 subj.) (Experimental): Ketamin-hameln (Ketaminhydrochlorid) 50mg/ml Ampullen; Hameln Pharma Plus GmbH; Sanova Pharma
  Dosis: 0.20mg/kg bodyweight bolus applied over 5 minutes (starting 15 minutes before PET measurement) and continuous infusion of 0.60mg/kg bodyweight applied over the course of 130 minutes.
  Pilot-study II is cross-over design!
  Interventions:
  Drug: (R,S)-ketamine (Pilot II) Other: PILOT Study II: PET1 Other: PILOT Study II: PET2
  Interventions: Drug: (R,S)-ketamine (Pilot II); Other: PILOT Study II: PET1; Other: PILOT Study II: PET2
- (R,S)-ketamine (Pilot Study I, 12 subj.) (Experimental): Ketamin-hameln (Ketaminhydrochlorid) 50mg/ml Ampullen; Hameln Pharma Plus GmbH; Sanova Pharma
  Dosis: 0.50mg/kg bodyweight i.v. over 40 Minutes (ending 5 minutes before PET measurement)
  Interventions:
  Drug: (R,S)-ketamine (Pilot I) Other: PILOT Study I: PET1 Other: PILOT Study I: PET2
  Interventions: Other: PILOT Study I: PET1; Other: PILOT Study I: PET2; Drug: (R,S)-ketamine (Pilot I)
- (R,S)-ketamine (Pilot Study III, 12 subj.) (Experimental): Ketamin-hameln (Ketaminhydrochlorid) 50mg/ml Ampullen; Hameln Pharma Plus GmbH; Sanova Pharma
  Dosis: 0.80mg/kg bodyweight i.v. over 50 Minutes
  Interventions:
  Drug: (R,S)-ketamine (Pilot III) Other: PILOT Study III: PET1 Other: PILOT Study III: PET2
  Interventions: Drug: (R,S)-ketamine (Pilot III); Other: PILOT Study III: PET1; Other: PILOT Study III: PET2

INTERVENTIONS:
Drug: (S)-ketamine (Main study) — Ketanest® S (Esketaminhydrochlorid) 5mg/ml and 25mg/ml ampoules; Actavis Italy S.P.A./Pfizer Corporation Austria GmbH
  Dosis: 0.25mg/kg bodyweight i.v. over 40 Minutes (ending 10 minutes before PET measurement)
  Other Names: Esketaminhydrochlorid
  Arms: (S)-ketamine
Drug: (S)-ketamine (Pilot II) — Ketanest® S (Esketaminhydrochlorid) 5mg/ml and 25mg/ml ampoules; Actavis Italy S.P.A./Pfizer Corporation Austria GmbH
  Dosis: 0.10mg/kg bodyweight i.v. bolus applied over 5 minutes (starting 15 minutes before PET measurement) and continuous infusion of 0.30mg/kg bodyweight i.v. applied over the course of 130 minutes.
  Other Names: Esketaminhydrochlorid
  Arms: (S)-ketamine (Pilot Study II, 5 subj.)
Drug: (R,S)-ketamine (Pilot II) — Ketamin-hameln (Ketaminhydrochlorid) 50mg/ml Ampullen; Hameln Pharma Plus GmbH; Sanova Pharma
  Dosis: 0.20mg/kg bodyweight i.v. bolus applied over 5 minutes (starting 15 minutes before PET measurement) and continuous infusion of 0.60mg/kg bodyweight applied i.v. over the course of 130 minutes.
  Other Names: Ketaminhydrochlorid
  Arms: (R,S)-ketamine (Pilot Study II, 5 subj.)
Drug: Placebo — 0.9% saline solution i.v. over 40 Minutes (ending 10 minutes before PET measurement)
  Arms: Placebo
Other: PILOT Study II: PET1 — [11C]DASB PET
  Arms: (R,S)-ketamine (Pilot Study II, 5 subj.); (S)-ketamine (Pilot Study II, 5 subj.)
Other: PILOT Study II: PET2 — [11C]DASB PET
  Arms: (R,S)-ketamine (Pilot Study II, 5 subj.); (S)-ketamine (Pilot Study II, 5 subj.)
Other: Main Study: PET1 — [11C]DASB PET
  Arms: (S)-ketamine; Placebo
Other: Main Study: PET2 — [11C]DASB PET
  Arms: (S)-ketamine; Placebo
Other: PILOT Study I: PET1 — [11C]DASB PET
  Arms: (R,S)-ketamine (Pilot Study I, 12 subj.)
Other: PILOT Study I: PET2 — [11C]DASB PET
  Arms: (R,S)-ketamine (Pilot Study I, 12 subj.)
Drug: (R,S)-ketamine (Pilot I) — Ketamin-hameln (Ketaminhydrochlorid) 50mg/ml Ampullen; Hameln Pharma Plus GmbH; Sanova Pharma
  Dosis: 0.50mg/kg bodyweight i.v. over 40 Minutes (ending 10 minutes before PET measurement)
  Other Names: Ketaminhydrochlorid
  Arms: (R,S)-ketamine (Pilot Study I, 12 subj.)
Drug: (R,S)-ketamine (Pilot III) — Ketamin-hameln (Ketaminhydrochlorid) 50mg/ml Ampullen; Hameln Pharma Plus GmbH; Sanova Pharma
  Dosis: 0.80mg/kg bodyweight i.v. over 50
  Other Names: Ketaminhydrochlorid
  Arms: (R,S)-ketamine (Pilot Study III, 12 subj.)
Other: PILOT Study III: PET1 — [11C]DASB PET
  Arms: (R,S)-ketamine (Pilot Study III, 12 subj.)
Other: PILOT Study III: PET2 — [11C]DASB PET
  Arms: (R,S)-ketamine (Pilot Study III, 12 subj.)

SUMMARY:
The study at hand is the first to investigate ketamine's SERT binding in humans, by utilizing the highly selective SERT radioligand [11C]DASB and positron emission tomography.

DETAILED DESCRIPTION:
Intravenous application of ketamine is currently dramatically gaining in significance as a rapid and highly effective antidepressant treatment option. Ketamine modulates various neurotransmitter systems, though the mechanisms responsible for its antidepressant effects remain unkownn. However, the serotonin transporter (SERT) presents a target of high interest due to the SERT's fundamental role in depression's pathophysiology as well as in antidepressant response. The study at hand is the first to investigate ketamine's SERT binding in humans, by utilizing the highly selective SERT radioligand [11C]DASB and positron emission tomography. Further, investigation of severely depressed patients provides the unique opportunity to establish the relationship between ketamine's SERT binding and its antidepressant efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years
* somatic health
* severe unipolar depression according to DSM-IV (SCID) und HAM-D (for patients)
* capable of giving informed consent
* negative pregnancy test (females)

Exclusion Criteria:

* severe somatic illness
* psychiatric disorder (for healthy controls)
* an axis I comorbidity other than MDD , other than anxiety symptoms (for patients)
* clinically relevant alterations in blood draw, ecg, and somatic testing
* substance dependency disorder
* intake of psychopharmacological medication in last 6 months
* first degree relative with Axis 1 disorder (for Pilot I study)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2016-05; Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Pilot Study II: (S)-ketamine SERT occupancy assessed with DASB binding potential (BP) | during PET/during 135 minutes of infusion
  Occupancy assessed using kinetic modeling
Pilot Study II: (R,S)-ketamine SERT occupancy assessed with DASB binding potential (BP) | during PET/during 135 minutes of infusion
  Occupancy assessed using kinetic modeling
Main Study: (S)-ketamine SERT occupancy assessed with DASB binding potential (BP) | during PET/starting 10 minutes afer 40 minutes of infusion
  Occupancy (%)=(1-BPND PET 2 (treatment) / BPND PET 1 (baseline)) x100
Pilot Study I: (R,S)-ketamine SERT occupancy assessed with DASB binding potential (BP) | during PET/starting 10 minutes afer 40 minutes of infusion
  Occupancy (%)=(1-BPND PET 2 (treatment) / BPND PET 1 (baseline)) x100
Pilot Study III: (R,S)-ketamine SERT occupancy assessed with DASB binding potential (BP) | during PET
  Occupancy (%)=(1-BPND PET 2 (treatment) / BPND PET 1 (baseline)) x100
Pilot Study III: resting state MRI | after PET 2
  changes to rsFC and rsfMRI after (R,S)-ketamine
Pilot Study III: MRS | after PET 2
  changes to Glutamate, GABA, and metabolites after (R,S)-ketami

SECONDARY OUTCOMES:
Change in Hamilton Depression Rating Scale Points | 2 hours after infusion to baseline
Change in Hamilton Depression Rating Scale Points | 1 day after infusion to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Lanzenberger, Prof., Principal Investigator — Department of Psychiatry and Psychotherapy, Medical University of Vienna
Locations (1):
- Department of Psychiatry and Psychotherapy, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Spies M, James GM, Berroteran-Infante N, Ibeschitz H, Kranz GS, Unterholzner J, Godbersen M, Gryglewski G, Hienert M, Jungwirth J, Pichler V, Reiter B, Silberbauer L, Winkler D, Mitterhauser M, Stimpfl T, Hacker M, Kasper S, Lanzenberger R. Assessment of Ketamine Binding of the Serotonin Transporter in Humans with Positron Emission Tomography. Int J Neuropsychopharmacol. 2018 Feb 1;21(2):145-153. doi: 10.1093/ijnp/pyx085. PMID 29045739